CLINICAL TRIAL: NCT02482766
Title: Efficacy of a New Technique -"IN-REC-SUR-E"- in Preterm Neonates With Respiratory Distress Syndrome During Non Invasive Ventilation: a Randomized Controlled Trial
Brief Title: Efficacy of a New Technique -"IN-REC-SUR-E"- in Preterm Neonates With RDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Ospedali Riuniti Ancona (Other); Careggi Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Centre for Neonatal Research and Education, Crawley, West Australia (Unknown); Monash University (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Giovanni VENTO, Associate Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prot. rs 25882/14
Record Dates: First submitted 2015-06-01; First posted 2015-06-26 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Respiratory Distress Syndrome; Hyaline Membrane Disease
MeSH Terms: conditions — Respiratory Distress Syndrome; Hyaline Membrane Disease | interventions — poractant alfa; Ventilators, Mechanical; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INRECSURE (Experimental): Infants in the INRECSURE arm will undergo the following approach: as soon as possible after the recruitment manoeuver (at CDP-Optimal) a dose of poractant alfa (Curosurf [Chiesi Farmaceutici, Parma, Italy]) of 200 mg/kg will be administered via a closed administration system in one-two aliquots (1-2 minutes). The tube position will be confirmed by auscultation. A temporary reduction of frequency may be necessary to increase the VT up to 2.5 ml/kg for improving the surfactant spreading.
  Interventions: Drug: Poractant alfa, 200 mg/kg; Device: Ventilator for High-frequency Oscillatory Ventilation (HFOV); Device: Nasal Continuous Positive Airway Pressure (nCPAP)
- INSURE (Active Comparator): Infants in the INSURE arm will undergo the following approach: after intubation, a dose of poractant alfa (Curosurf [Chiesi Farmaceutici, Parma, Italy]) of 200 mg/kg will be administered via a closed administration system in one-two aliquots (1-2 minutes). The tube position will be confirmed by auscultation. During surfactant administration, infants will be manually ventilated to facilitate surfactant distribution.
  Interventions: Drug: Poractant alfa, 200 mg/kg; Device: Nasal Continuous Positive Airway Pressure (nCPAP)

INTERVENTIONS:
Drug: Poractant alfa, 200 mg/kg — Endotracheal Surfactant administration
  Other Names: Curosurf-Chiesi Farmaceutici, Parma, Italy
Device: Ventilator for High-frequency Oscillatory Ventilation (HFOV) — This device will be used to perform an HFOV recruitment maneuver before surfactant administration
  Arms: INRECSURE
Device: Nasal Continuous Positive Airway Pressure (nCPAP) — After surfactant administration, the babies will be extubated within 30 minutes and will receive nCPAP (6-8 cm H2O)

SUMMARY:
The primary hypothesis of this study is reduction in need of mechanical ventilation in the first 72 hours of life (excluding the transient tracheal intubation performed for surfactant administration and the mechanical ventilation for lung recruitment) in spontaneously breathing infants born at 24+0-27+6 weeks' gestation and failing nCPAP during the first 24 hours of life who received an HFOV recruitment maneuver (IN-REC-SUR-E) compared to no recruitment maneuver (IN-SUR-E) just prior to surfactant administration followed by prompt extubation.

DETAILED DESCRIPTION:
EFFICACY OF A NEW TECHNIQUE -"IN-REC-SUR-E"- IN PRETERM NEONATES WITH RESPIRATORY DISTRESS SYNDROME DURING NON INVASIVE VENTILATION: A RANDOMIZED CONTROLLED TRIAL

BACKGROUND The initial stabilization on Continuous Positive Airway Pressure (CPAP) and provision of rescue surfactant only when necessary is at least as beneficial and quite possibly preferred over the standard therapy of intubation of all infants at risk in the delivery room and subsequent support with mechanical ventilation (2-4). The percentage of CPAP failure in the newborns of 25-28 weeks' gestation is 45 % (30/66) in the Australian experience (5), higher than that reported by Ammari et al. (25 %) (6) and similar to that reported by De Jaegere et al. (50 %) (7) and in the COIN trial (46 %) (2). As a potential alternative, the INSURE (INtubate, SURfactant, Extubate) approach (8) is very attractive. Recently, several studies have investigated the effectiveness of the association between non-invasive ventilation and surfactant, administered by transient intubation (INSURE), showing that it is effective in preventing the need for mechanical ventilation. Although beneficial in clinical practice, the INSURE method cannot be universally applied to all preterm neonates with Respiratory Distress Syndrome (RDS) and is unsuccessful in a particular section of this population. The INSURE failure rate recently reported in preterm infants of different gestational age widely ranges from 19 % to 69 % (10, 11). Unfortunately, no randomized controlled trials have directly evaluated the efficacy of INSURE in extremely preterm neonates (<28 weeks gestation) (8). Nevertheless, the data of the "Sustained Lung Inflation (SLI) study" (14) recently conducted on infants with GA 25+0- 28+6 weeks showed that nasal CPAP failure and need for Mechanical Ventilation (MV) at 72 hours of life was 53 % in the SLI group and 65 % in the control group (only nasal CPAP). In this study surfactant was preferably administered with the INSURE approach at a Fraction of Inspired Oxygen (FiO2) threshold of 0.40 and then it could be reasonably argued that at least 50 % of 25-28 weeks' gestation infants, even if receiving a SLI maneuver and the INSURE treatment for CPAP failure, undergoes mechanical ventilation in the first 72 hours of life for unsuccessful INSURE. One of the possible mechanisms responsible for the unsuccessful INSURE, requiring subsequent re-intubation and mechanical ventilation is the inability of the preterm lung with RDS of achieving and maintaining an "optimal" Functional Residual Capacity (FRC). Prophylactic or early rescue surfactant administration before alveolar recruitment probably results in an uneven surfactant distribution to already open alveoli thus resulting in poor clinical response to the first surfactant treatment. We, therefore, seek to compare the application of a recruitment manoeuver - in High-Frequency Oscillatory Ventilation (HFOV) modality - just before the surfactant administration, followed by rapid extubation (INtubate-RECruited-SURfactant-Extubation: IN-REC-SUR-E) with INSURE alone in spontaneously breathing preterm infants requiring nasal CPAP as initial respiratory support and reaching pre-defined CPAP failure criteria, for evaluating its effectiveness in decreasing the need of MV and improving respiratory outcome.

Study design This will be an unblinded multi-center randomized trial of IN-REC-SUR-E vs. IN-SUR-E in infants born at 24+0-27+6 weeks' gestation.

Sample size The investigators hypothesized that a recruitment manoeuver (in HFOV modality) before surfactant administration might decrease of the need of subsequent mechanical ventilation during the first 72 hours of life from 50 % (2, 5, 7) to 30 %. The investigators calculated that 103 newborns must be enrolled in each group to detect this difference as statistically significant with 80 % power at 0.05 level.

Randomisation Infants at each unit will be block (1st block: gestational age from 24+0 to 25+6 weeks; 2nd block: gestational age from 26+0 to 27+6 weeks) randomly assigned to a treatment group using automatically generated sealed envelopes which will be prepared at Policlinico A. Gemelli Hospital in Rome and then distributed to participating centers. Permutated block randomization with 1:1 randomization between the two arms will be used.

Blinding The study will not be blinded, and the staff performing the study also will take care of the infants later on. However, the decision to start mechanical ventilation will be made by clinicians other than the investigators and, moreover, parents, nurses involved in patient care and researchers assessing study end-points will be blinded to the nature of the study treatments. To minimize bias, strict criteria and definitions will be maintained during the trial.

Management in the Delivery Room Positive pressure with a neonatal mask and a T-piece system (Neopuff Infant Resuscitator, Fisher and Paykel, Auckland, New Zealand) will be used to stabilize newborns after birth. All the neonates will receive one (or two) SLI manoeuver(s) (25 cmH2O for 10-15 seconds) (14) and will be transferred to the Neonatal Intensive Care Unit (NICU) in nasal CPAP (6 cmH2O). Infants will start mechanical ventilation in agreement with the American Academy of Paediatrics guidelines on neonatal resuscitation (16). In this latter case the babies will be excluded from the study (see exclusion criteria section, page 4).

CPAP Failure Criteria In the NICU, nasal CPAP will be given through nasal prongs/mask using the standard method of the single centre (ventilator, flow-dependent system) with an initial pressure of 6 to 7 cmH2O, in all infants. CPAP failure is defined if they met any of the following criteria: FiO2 ≥ 0.30 on nasal CPAP (17) to maintain pulse oximetry (SpO2) 87-94 %(18) for at least 30 minutes unless rapid clinical deterioration occurred, respiratory acidosis defined as pCO2 > 65 mmHg (8.5 kPa) and pH < 7.20 on arterial or capillary blood gas sample, apnea defined as >4 episodes of apnea per hour or >2 episodes of apnea per hour when ventilation with bag and mask will be required.

HFOV Recruitment manoeuver Infants in the IN-REC-SUR-E group will undergo the following approach: after intubation, HFOV will be delivered with the ventilator available in each NICU. The following initial ventilator setting will be advocated: Continuous Distending Pressure (CDP): 8cmH2O; Frequency: 10-15 Hz; Delta P: 15 cmH2O or Amplitude 30 % eventually increased - chest to be "visibly vibrating "-; I:E 1:2. Delta P (or amplitude) first and/or frequency subsequently will be adjusted to achieve a Tidal Volume (VT) of 1,5-2 ml/kg and/or to maintain the transcutaneous partial carbon dioxide pressure (TcPCO2) between 40 and 60 mmHg (5.3 and 8.0 kPa). The infants will be subjected to an open lung ventilation strategy aiming to recruit and stabilize the majority of collapsed alveoli/sacculi, using oxygenation as an indirect parameter for lung volume. Optimal recruitment is defined as adequate oxygenation using a FiO2 of 0.25 or less. Starting at 8 cmH2O, the CDP will be increased stepwise (2 cmH2O every 2-3 minutes) as long as SpO2 improves. The FiO2 will be reduced stepwise, keeping SpO2 within the target range (87-94 %). The recruitment procedure will be stopped if oxygenation no longer improves or if the FiO2 is equal to or less than 0.25. The corresponding CDP will be called the opening pressure (CDPO). Next, the CDP will be reduced stepwise (1-2 cmH2O every 2-3 minutes) until the SpO2 deteriorates (of at least 2-3 points). The corresponding CDP will be called the closing pressure (CDPC). After a second recruitment manoeuver at CDPO for 2 minutes, the optimal CDP (CDPOPT) will be set 2 cmH2O above the CDPC for at least 3 minutes (19). A chest radiograph at this point is advised.

Surfactant Treatment

Infants in the IN-REC-SUR-E arm will undergo the following approach: as soon as possible after the recruitment manoeuver (at CDPOPT) a dose of poractant alfa (Curosurf [Chiesi Farmaceutici, Parma, Italy]) of 200 mg/kg will be administered via a closed administration system in one-two aliquots (1-2 minutes). The tube position will be confirmed by auscultation. A temporary reduction of frequency may be necessary to increase the VT up to 2.5 ml/kg for improving the surfactant spreading.

Infants in the IN-SUR-E arm will undergo the following approach: after intubation, a dose of poractant alfa (Curosurf [Chiesi Farmaceutici, Parma, Italy]) of 200 mg/kg will be administered via a closed administration system in one-two aliquots (1-2 minutes). The tube position will be confirmed by auscultation. During surfactant administration, infants will be manually ventilated to facilitate surfactant distribution. If necessary, mechanical ventilation with a peak inspiratory pressure (PIP) of 20-22 cmH2O, a Positive End-Expiratory Pressure (PEEP) of 5-6 cmH2O and a respiratory rate of 30-40 breaths/min will be subsequently started to achieve a VT of 4-6 ml/kg and/or to maintain the transcutaneous partial carbon dioxide pressure (TcPCO2) between 40 and 60 mmHg (5.3 and 8.0 kPa).

After surfactant administration, the babies of both groups will be extubated within 30 minutes (if satisfactory respiratory drive is present) and will receive nasal CPAP (6-8 cmH2O) (20). In case of insufficient respiratory drive, CDP (in the babies of IN-REC-SUR-E arm) or PIP (in the IN-SUR-E arm) will be reduced until spontaneous respiratory activity is restored. Maintaining a FiO2 < 0.30 to obtain SpO2 values in the desired range (87-94 %) will drive the eventual reduction in the level of CPAP in the following days. The decision as to whether to begin Bi-level Positive Airway Pressure (BiPAP) or nasal-Intermittent Mandatory Ventilation (N-IMV) to prevent the need for re-intubation in infants of both groups will be up to the neonatologist on duty, and will be considered in the final analysis.

Infants of both groups can receive a subsequent dose of surfactant (100 mg/kg of poractant alfa) using the same method (INSURE or INRECSURE) if they meet the CPAP failure criteria again during the following 12 to 24 hours.

Data collection All collected data can be obtained from the clinical records. They will be reported in electronic data sheets designed for this study.

Statistical analysis The primary efficacy analysis will be conducted on an intention to treat basis. Clinical characteristics of infants in the "IN-REC-SUR-E" and "IN-SUR-E" groups will be described using mean values and standard deviation, median value and range, or rate and percentage. Univariate statistical analysis will be performed using the Student "t" test for parametric continuous variables, the Wilcoxon rank-sum test for non-parametric continuous variables, and Fisher's exact test for categorical variables. A p <0.05 will be considered statistically significant. Then, "IN-REC-SUR-E" treatment and clinical characteristics which are most likely associated with the need for mechanical ventilation (gestational age, birth weight, antenatal steroids, CRIB score) will be included in multiple logistic regression analysis to assess their independent role in predicting "IN-REC-SUR-E" success or failure. Effect estimates will be expressed as relative risk (RR) with profile likelihood-based 95 % confidence limits.

An interim analysis is planned when 50 infants will be enrolled in each arm. Duration of study: 1 year

QUALITY CONTROL AND QUALITY ASSURANCE PROCEDURES Compliance to protocol Compliance will be defined as full adherence to protocol. Compliance with the protocol will be ensured by a number of procedures as described below.

Site set-up Local principal investigators are required to participate in preparatory meetings in which details of study protocol, data collection, "IN-REC-SUR-E" and "IN-SUR-E" procedures will be accurately discussed. All centers will receive detailed written instruction on web based data recording, and, to solve possible difficulties, it will be possible to contact the Clinical Trials Coordinating Center. Moreover, it has been ascertained that "IN-REC-SUR-E" procedure is followed similarly in all participating centers.

ELIGIBILITY:
Inclusion Criteria:

1. In-Born at 24+0-27+6 (and)
2. Spontaneously breathing at birth but requiring respiratory support (CPAP or O2) at 5' of life (and)
3. Parental consent has been obtained (and)
4. Failing nCPAP during the first 24 hours of life

Exclusion Criteria:

1. Severe birth asphyxia or a 5-minute Apgar score <3
2. Endotracheal intubation in the delivery room for resuscitation or insufficient respiratory drive according to AAP guidelines16
3. Prolonged PROM > 3 weeks
4. Presence of major congenital malformations
5. Hydrops fetalis
6. Inherited disorders of metabolism

Ages: 24 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2015-11; Primary Completion 2018-09 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Need for mechanical ventilation within the first 3 days of life and therefore we consider IN-REC-SUR-E a success if mechanical ventilation is not required and a failure if the infant needs mechanical ventilation in the first 72 hours. | First 72 hours of life

SECONDARY OUTCOMES:
Duration of NCPAP | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Duration of conventional mechanical ventilation | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Duration of High-frequency oscillatory ventilation (HFOV) | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Duration of O2-therapy | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Duration of hospitalization | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Number of doses of surfactant | First 72 hours of life
Occurrence of BPD (mild, moderate and severe forms) | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Time to be out of any respiratory support | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks

OTHER OUTCOMES:
Air leaks | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  "Mono or bilateral pneumothorax" ; "Pulmonary interstitial Emphysema"
Pulmonary hemorrage | First 72 hours of life
  Sudden onset of overt bleeding or frank evidence of blood in the airway, leading to acute respiratory distress or respiratory failure, with diffuse, bilateral pulmonary infiltrates on chest radiograph.
PDA and need of surgical closure | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Hour(s) of administration of surfactant dose(s) | First 72 hours of life
3°- 4° IVH | First week of life
PVL | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
>2° ROP | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
NEC | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Sepsis | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Sepsis is defined as a positive blood culture or suggestive clinical and laboratory findings leading to treatment with antibiotics for at least 7 days despite absence of a positive blood culture.
Lenght of stay in NICU | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Use of systemic postnatal steroids | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks
  Number of cycles of postnatal steroids i.v.: "None", "1", "> 1 cycle"
Mortality | Participants will be followed for the duration of hospital stay, an expected average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Vento, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (33):
- Italy (33):
  - Ospedale Salesi, Ancona, AN
  - Ospedale Di Venere, Bari, BA
  - Ospedale Maggiore, Bologna, BO
  - Fondazione Poliambulanza, Brescia, BS
  - Ospedale di Bolzano, Bolzano, BZ
  - Pineta Grande, Caserta, CE
  - S. Sebastiano e S. Anna, Caserta, CE
  - Azienda Ospedaliera di Cosenza, Cosenza, CS
  - AOU Policlinico Vittorio Emanuele- Presidio Ospedaliero Gaspare Rodolico, Catania, CT
  - Ospedale Nuovo Garibaldi-Nesima, Catania, CT
  - Ospedale Vito Fazzi, Lecce, LE
  - Ospedale Barone Romeo, Patti, ME
  - Ospedale san Pietro Fatebenefratelli, Rome, RM
  - Ospedale San Bortolo, Vicenza, VI
  - SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Universitaria Ferrara, Ferrara
  - Careggi, Florence
  - Ospedali Riuniti, Foggia
  - Ospedale San Salvatore, L’Aquila
  - Carlo Poma, Mantova
  - Università degli studi di Messina A.O.U. Policlinico G. Martino, Messina
  - Mangiagalli, Milan
  - Ospedale Niguarda, Milan
  - A.O.U. di Modena Policlinico, Modena
  - S. Gerardo, Monza
  - Ospedale Maggiore, Novara
  - Arnas Civico di Palermo, Palermo
  - A.O. Bianchi-Melacrino-Morelli, Reggio Calabria
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fatebenefratelli-Isola Tiberina, Roma
  - Policlinico Gemelli-Università Cattolica S. Cuore, Rome
  - A.O. Treviso Ospedale Cà Foncello, Treviso
  - Belcolle, Viterbo

REFERENCES:
- [Result] Van Marter LJ, Allred EN, Pagano M, Sanocka U, Parad R, Moore M, Susser M, Paneth N, Leviton A. Do clinical markers of barotrauma and oxygen toxicity explain interhospital variation in rates of chronic lung disease? The Neonatology Committee for the Developmental Network. Pediatrics. 2000 Jun;105(6):1194-201. doi: 10.1542/peds.105.6.1194. PMID 10835057
- [Result] Morley CJ, Davis PG, Doyle LW, Brion LP, Hascoet JM, Carlin JB; COIN Trial Investigators. Nasal CPAP or intubation at birth for very preterm infants. N Engl J Med. 2008 Feb 14;358(7):700-8. doi: 10.1056/NEJMoa072788. PMID 18272893
- [Result] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Result] Dunn MS, Kaempf J, de Klerk A, de Klerk R, Reilly M, Howard D, Ferrelli K, O'Conor J, Soll RF; Vermont Oxford Network DRM Study Group. Randomized trial comparing 3 approaches to the initial respiratory management of preterm neonates. Pediatrics. 2011 Nov;128(5):e1069-76. doi: 10.1542/peds.2010-3848. Epub 2011 Oct 24. PMID 22025591
- [Result] Dargaville PA, Aiyappan A, De Paoli AG, Dalton RG, Kuschel CA, Kamlin CO, Orsini F, Carlin JB, Davis PG. Continuous positive airway pressure failure in preterm infants: incidence, predictors and consequences. Neonatology. 2013;104(1):8-14. doi: 10.1159/000346460. Epub 2013 Apr 4. PMID 23595061
- [Result] Ammari A, Suri M, Milisavljevic V, Sahni R, Bateman D, Sanocka U, Ruzal-Shapiro C, Wung JT, Polin RA. Variables associated with the early failure of nasal CPAP in very low birth weight infants. J Pediatr. 2005 Sep;147(3):341-7. doi: 10.1016/j.jpeds.2005.04.062. PMID 16182673
- [Result] De Jaegere AP, van der Lee JH, Cante C, van Kaam AH. Early prediction of nasal continuous positive airway pressure failure in preterm infants less than 30 weeks gestation. Acta Paediatr. 2012 Apr;101(4):374-9. doi: 10.1111/j.1651-2227.2011.02558.x. Epub 2012 Jan 9. PMID 22150698
- [Result] Stevens TP, Harrington EW, Blennow M, Soll RF. Early surfactant administration with brief ventilation vs. selective surfactant and continued mechanical ventilation for preterm infants with or at risk for respiratory distress syndrome. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD003063. doi: 10.1002/14651858.CD003063.pub3. PMID 17943779
- [Result] Sandri F, Plavka R, Ancora G, Simeoni U, Stranak Z, Martinelli S, Mosca F, Nona J, Thomson M, Verder H, Fabbri L, Halliday H; CURPAP Study Group. Prophylactic or early selective surfactant combined with nCPAP in very preterm infants. Pediatrics. 2010 Jun;125(6):e1402-9. doi: 10.1542/peds.2009-2131. Epub 2010 May 3. PMID 20439601
- [Result] Brix N, Sellmer A, Jensen MS, Pedersen LV, Henriksen TB. Predictors for an unsuccessful INtubation-SURfactant-Extubation procedure: a cohort study. BMC Pediatr. 2014 Jun 19;14:155. doi: 10.1186/1471-2431-14-155. PMID 24947477
- [Result] Lakkundi A, Wright I, de Waal K. Transitional hemodynamics in preterm infants with a respiratory management strategy directed at avoidance of mechanical ventilation. Early Hum Dev. 2014 Aug;90(8):409-12. doi: 10.1016/j.earlhumdev.2014.04.017. Epub 2014 Jun 5. PMID 24951077
- [Result] Dani C, Corsini I, Bertini G, Fontanelli G, Pratesi S, Rubaltelli FF. The INSURE method in preterm infants of less than 30 weeks' gestation. J Matern Fetal Neonatal Med. 2010 Sep;23(9):1024-9. doi: 10.3109/14767050903572174. PMID 20180736
- [Result] Cherif A, Hachani C, Khrouf N. Risk factors of the failure of surfactant treatment by transient intubation during nasal continuous positive airway pressure in preterm infants. Am J Perinatol. 2008 Nov;25(10):647-52. doi: 10.1055/s-0028-1090590. Epub 2008 Oct 7. PMID 18841536
- [Result] Lista G, Boni L, Scopesi F, Mosca F, Trevisanuto D, Messner H, Vento G, Magaldi R, Del Vecchio A, Agosti M, Gizzi C, Sandri F, Biban P, Bellettato M, Gazzolo D, Boldrini A, Dani C; SLI Trial Investigators. Sustained lung inflation at birth for preterm infants: a randomized clinical trial. Pediatrics. 2015 Feb;135(2):e457-64. doi: 10.1542/peds.2014-1692. PMID 25624390
- [Result] Krause MF, Jakel C, Haberstroh J, Schulte-Monting J, Leititis JU, Orlowska-Volk M. Alveolar recruitment promotes homogeneous surfactant distribution in a piglet model of lung injury. Pediatr Res. 2001 Jul;50(1):34-43. doi: 10.1203/00006450-200107000-00009. PMID 11420416
- [Result] Perlman JM, Wyllie J, Kattwinkel J, Atkins DL, Chameides L, Goldsmith JP, Guinsburg R, Hazinski MF, Morley C, Richmond S, Simon WM, Singhal N, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Neonatal resuscitation: 2010 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Pediatrics. 2010 Nov;126(5):e1319-44. doi: 10.1542/peds.2010-2972B. Epub 2010 Oct 18. No abstract available. PMID 20956431
- [Result] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Halliday HL; European Association of Perinatal Medicine. European consensus guidelines on the management of neonatal respiratory distress syndrome in preterm infants--2013 update. Neonatology. 2013;103(4):353-68. doi: 10.1159/000349928. Epub 2013 May 31. PMID 23736015
- [Result] Sola A, Golombek SG, Montes Bueno MT, Lemus-Varela L, Zuluaga C, Dominguez F, Baquero H, Young Sarmiento AE, Natta D, Rodriguez Perez JM, Deulofeut R, Quiroga A, Flores GL, Morgues M, Perez AG, Van Overmeire B, van Bel F. Safe oxygen saturation targeting and monitoring in preterm infants: can we avoid hypoxia and hyperoxia? Acta Paediatr. 2014 Oct;103(10):1009-18. doi: 10.1111/apa.12692. Epub 2014 Jul 28. PMID 24838096
- [Result] De Jaegere A, van Veenendaal MB, Michiels A, van Kaam AH. Lung recruitment using oxygenation during open lung high-frequency ventilation in preterm infants. Am J Respir Crit Care Med. 2006 Sep 15;174(6):639-45. doi: 10.1164/rccm.200603-351OC. Epub 2006 Jun 8. PMID 16763218
- [Result] Buzzella B, Claure N, D'Ugard C, Bancalari E. A randomized controlled trial of two nasal continuous positive airway pressure levels after extubation in preterm infants. J Pediatr. 2014 Jan;164(1):46-51. doi: 10.1016/j.jpeds.2013.08.040. Epub 2013 Oct 1. PMID 24094879
- [Result] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Result] Parry G, Tucker J, Tarnow-Mordi W; UK Neonatal Staffing Study Collaborative Group. CRIB II: an update of the clinical risk index for babies score. Lancet. 2003 May 24;361(9371):1789-91. doi: 10.1016/S0140-6736(03)13397-1. PMID 12781540
- [Result] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Result] de Vries LS, Eken P, Dubowitz LM. The spectrum of leukomalacia using cranial ultrasound. Behav Brain Res. 1992 Jul 31;49(1):1-6. doi: 10.1016/s0166-4328(05)80189-5. PMID 1388792
- [Result] International Committee for the Classification of Retinopathy of Prematurity. The International Classification of Retinopathy of Prematurity revisited. Arch Ophthalmol. 2005 Jul;123(7):991-9. doi: 10.1001/archopht.123.7.991. PMID 16009843
- [Result] Bell MJ, Ternberg JL, Feigin RD, Keating JP, Marshall R, Barton L, Brotherton T. Neonatal necrotizing enterocolitis. Therapeutic decisions based upon clinical staging. Ann Surg. 1978 Jan;187(1):1-7. doi: 10.1097/00000658-197801000-00001. PMID 413500
- [Derived] Vento G, Ventura ML, Pastorino R, van Kaam AH, Carnielli V, Cools F, Dani C, Mosca F, Polglase G, Tagliabue P, Boni L, Cota F, Tana M, Tirone C, Aurilia C, Lio A, Costa S, D'Andrea V, Lucente M, Nigro G, Giordano L, Roma V, Villani PE, Fusco FP, Fasolato V, Colnaghi MR, Matassa PG, Vendettuoli V, Poggi C, Del Vecchio A, Petrillo F, Betta P, Mattia C, Garani G, Solinas A, Gitto E, Salvo V, Gargano G, Balestri E, Sandri F, Mescoli G, Martinelli S, Ilardi L, Ciarmoli E, Di Fabio S, Maranella E, Grassia C, Ausanio G, Rossi V, Motta A, Tina LG, Maiolo K, Nobile S, Messner H, Staffler A, Ferrero F, Stasi I, Pieragostini L, Mondello I, Haass C, Consigli C, Vedovato S, Grison A, Maffei G, Presta G, Perniola R, Vitaliti M, Re MP, De Curtis M, Cardilli V, Lago P, Tormena F, Orfeo L, Gizzi C, Massenzi L, Gazzolo D, Strozzi MCM, Bottino R, Pontiggia F, Berardi A, Guidotti I, Cacace C, Meli V, Quartulli L, Scorrano A, Casati A, Grappone L, Pillow JJ. Lung recruitment before surfactant administration in extremely preterm neonates with respiratory distress syndrome (IN-REC-SUR-E): a randomised, unblinded, controlled trial. Lancet Respir Med. 2021 Feb;9(2):159-166. doi: 10.1016/S2213-2600(20)30179-X. Epub 2020 Jul 17. PMID 32687801
- [Derived] Vento G, Pastorino R, Boni L, Cota F, Carnielli V, Cools F, Dani C, Mosca F, Pillow J, Polglase G, Tagliabue P, van Kaam AH, Ventura ML, Tana M, Tirone C, Aurilia C, Lio A, Ricci C, Gambacorta A, Consigli C, D'Onofrio D, Gizzi C, Massenzi L, Cardilli V, Casati A, Bottino R, Pontiggia F, Ciarmoli E, Martinelli S, Ilardi L, Colnaghi M, Matassa PG, Vendettuoli V, Villani P, Fusco F, Gazzolo D, Ricotti A, Ferrero F, Stasi I, Magaldi R, Maffei G, Presta G, Perniola R, Messina F, Montesano G, Poggi C, Giordano L, Roma E, Grassia C, Ausanio G, Sandri F, Mescoli G, Giura F, Garani G, Solinas A, Lucente M, Nigro G, Del Vecchio A, Petrillo F, Orfeo L, Grappone L, Quartulli L, Scorrano A, Messner H, Staffler A, Gargano G, Balestri E, Nobile S, Cacace C, Meli V, Dallaglio S, Pasqua B, Mattia L, Gitto E, Vitaliti M, Re MP, Vedovato S, Grison A, Berardi A, Torcetta F, Guidotti I, di Fabio S, Maranella E, Mondello I, Visentin S, Tormena F. Efficacy of a new technique - INtubate-RECruit-SURfactant-Extubate - "IN-REC-SUR-E" - in preterm neonates with respiratory distress syndrome: study protocol for a randomized controlled trial. Trials. 2016 Aug 18;17:414. doi: 10.1186/s13063-016-1498-7. PMID 27538798